CLINICAL TRIAL: NCT04237480
Title: Influence of Kidney Performance and Magnesium on the Biomarkers of Vitamin D
Brief Title: Influence of Kidney Performance and Magnesium on Formation of (OH)2-vitamin D3
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00923
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hydroxylase Deficiency
Keywords: vitamin D; 1-alpha hydroxylase; magnesium; renal insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum value 1,25(OH)2 vitamin D — statistical evaluation of the serum values
  Other Names: serum value 25(OH) vitamin D; serum value magnesium; serum value creatinine

SUMMARY:
Retrospective database analysis. The target values are the serum values of 25(OH)D, of 1,25(OH)2D, of magnesium and creatinine as well as age and sex of the patients. The laboratory values of the years 2017 and 2018 are included. There are no additional measurements on patients.

DETAILED DESCRIPTION:
The laboratory values of the years 2017 and 2018 are included. All laboratory results to be evaluated originate from Medics Labor in Bern. We expect about 50'000 data sets. It is impossible for the study team to draw conclusions about the patients or the senders.

ELIGIBILITY:
Inclusion Criteria:

* all data sets available

Exclusion Criteria:

* a declaration from the patient that his laboratory values may not be included in an evaluation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: no restriction
Sampling Method: Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
correlation of serum values of 1,25(OH)2 vitamin D with estimated glomerular filtration rate | 2017 - 2018
  statistical evaluation of serum values
correlation of serum values of 1,25(OH)2 vitamin D with magnesium | 2017 - 2018
  statistical evaluation of serum values

IPD SHARING:
Plan to Share IPD: No